CLINICAL TRIAL: NCT01887444
Title: The Benefit of Using the Lactobacillus Reuteri Probiotic as a Supplement in the Treatment of Newborn Colic
Brief Title: Lactobacillus Reuteri Supplementation in the Treatment of Infantile Colic
Acronym: PROBIOC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Never started
Sponsor: BioGaia AB (Industry)
Collaborators: CRC CHI Creteil France (Other Government); Association Clinique Thérapeutique Infantile du val de Marne (Other); Hopital Universitaire Robert-Debre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013-A00163-42
Record Dates: First submitted 2013-06-20; First posted 2013-06-26 (Estimated); Last update posted 2021-02-04 (Actual); Status verified 2015-09

CONDITIONS: Infantile Colic
Keywords: Pediatric Gastroenterology; Probiotics; Lactobacillus reuteri
MeSH Terms: conditions — Colic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lactobacillus reteuri (Experimental): Dietary Supplement: Lactobacillus reuteri DSM17938 probiotic 2 x 10(8) CFU/day 21 days
  Interventions: Dietary Supplement: Lactobacillus reuteri DSM17938 probiotic
- Placebo (Placebo Comparator): Other: Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus reuteri DSM17938 probiotic — Drops suitable for infants. 2 X 5 drops / day will be issued, corresponding to 2.108 CFU Lactobacillus reuteri living DSM17938. The probiotic is contained in a lipid emulsion.
  Arms: Lactobacillus reteuri
Other: Placebo — Drops suitable for infants. 2 X 5 drops / day will be issued, corresponding to the lipid emulsion without probiotics.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of the oral administration of Lactobacillus reuteri in treating infantile colic as defined by the Rome III criteria. Forty breastfed infants aged from 29 days to 3 months will be enrolled and blinded randomized to receive orally L.reuteri or placebo. The rate of responders (reduction of daily crying time >50% compared to the baseline) will be assessed at day 7, day 14 and day 21 in both groups. The average daily crying time as well as the associated digestive symptoms will also be analyzed.

DETAILED DESCRIPTION:
NOTE: The study never started.

ELIGIBILITY:
Inclusion Criteria:

1. Exclusively breastfed Infants
2. Infant aged of 29 days to 3 months
3. With a diagnosis of infantile colic as defined by the Rome III criteria
4. Birth at term and eutrophic (weight, height, head circumference)
5. Apgar score> 7 at 5 minutes
6. Consent to the study signed by the two parents.
7. Availability during the study period

Exclusion Criteria:

1. Associated severe chronic disease
2. Acute infectious disease
3. Personal or family first degree history of allergy to milk proteins
4. Several infants of the same family from a multiple pregnancy
5. Infants who received antibiotics one week prior to randomization
6. Infants who received probiotics one week prior to randomization
7. Mother who received antibiotics 1 week before randomization
8. Regular consumption of probiotics by the mother 1 week before randomization
9. Infants-included in another clinical study
10. Lack of insurance coverage by the french social security
11. Non exclusively breastfed infants

Ages: 29 Days to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2014-05 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
The responder rate (infants for whom daily crying time decreases by 50% compared to baseline, D0) at D7 in the probiotic group compared to placebo. The daily crying time will be sound recorded during 24 hours at D0 and D7.and expressed in minutes. | day 7

SECONDARY OUTCOMES:
The responders rates at D14 and D21 in the probiotic group compared to the placebo group. | Day 14 and day 21

OTHER OUTCOMES:
The average duration of crying in the probiotic group compared with the placebo group at D7, D14 and D21. | Day 7, 14 and 21
Gastrointestinal symptoms (constipation, diarrhea, flatulence) evaluated at each visit required by the protocol | day 7, 14 and 21

CONTACTS AND LOCATIONS:
Overall Officials: Marc Bellaiche, MD, Principal Investigator — Hopital Universitaire Robert-Debre
Locations (1):
- CRC CHIC and ACTIV, Créteil, France